CLINICAL TRIAL: NCT05018780
Title: Immediate and Long Term Effects of Muscle Energy Techniques and Sacral Manipulation on Pain, Functional Disability and Quality of Life in Patients With Sacroiliac Joint Dysfunction: A Randomized Clinical Trial
Brief Title: Muscle Energy Techniques and Sacral Manipulation on Pain, Functional Disability and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/885/2021
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2021-12

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroilitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study will be single and assessor blinded. Participants will be masked about other groups but they will know what treatment they will be receiving or what exercises they will be doing. Principal investigator would also not be masked or blinded because investigator would be applying the techniques on participants of both group. So participant and and principal investigator cannot be blinded. Only assessor will be blinded and he will take outcome measures without knowing the problem and treatment techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Post isometric relaxation: Patient will perform isometrics on piriformis, iliopsoas and erector spinae muscles one by one. Each isometric contraction will be held for 10 seconds and than participants will be asked to relax the contraction with an exhalation. This will be repeated five times in one session.
  - Routine physical therapy including TENS, Hot pack and strengthening exercises will also be delivered along with Muscle Energy Technique.
  Interventions: Other: Muscle Energy Technique
- Sacral Manipulation (Experimental): * To manipulate an iliac anterior rotation displacement sacroiliac joint dysfunction and to restore posterior rotation of the ilium, participant will be positioned in side lying. Therapist will place one hand at Anterior superior iliac supine (ASIS) and the other at Ischial tuberosity. A quick thrust will be applied and ASIS will be pushed posteriorly while Ischial tberosity anteriorly. This will be maintained for 10 to 30 seconds.
  * To manipulate an iliac posterior rotation displacement sacroiliac joint dysfunction and to restore anterior rotation of the ilium, participant will be in prone position. One hand of therapist will be at Posterior superior iliac supine (PSIS) and the other one at pubic rami. A quick thrust will be delivered and PSIS will be moved anteriorly while pubic rami posteriorly. This will be maintained for 10 to 30 seconds.
  * Routine physical therapy including TENS, Hot pack and strengthening exercises will also be delivered along with Sacral Manipulation.
  Interventions: Other: Sacral Manipulation

INTERVENTIONS:
Other: Muscle Energy Technique — Post isometric relaxation: Patient will be asked to perform isometrics on piriformis, iliopsoas and erector spinae muscles one by one. Each isometric contraction will be held for 10 seconds. After 10 seconds, contraction will be released with an exhalation. These contractions will be repeated for 5 times in one session.
  Routine physical therapy including TENS, Hot pack and strengthening exercises will also be delivered along with Muscle Energy Technique.
  Arms: Muscle Energy Technique
Other: Sacral Manipulation — * To manipulate an iliac anterior rotation displacement sacroiliac joint dysfunction and to restore posterior rotation of the ilium, participant will be positioned in side lying. Therapist will place one hand at Anterior superior iliac supine (ASIS) and the other at Ischial tuberosity. A quick thrust will be applied and ASIS will be pushed posteriorly while Ischial tberosity anteriorly. This will be maintained for 10 to 30 seconds.
  * To manipulate an iliac posterior rotation displacement sacroiliac joint dysfunction and to restore anterior rotation of the ilium, participant will be in prone position. One hand of therapist will be at Posterior superior iliac supine (PSIS) and the other one at pubic rami. A quick thrust will be delivered and PSIS will be moved anteriorly while pubic rami posteriorly. This will be maintained for 10 to 30 seconds.
  * Routine physical therapy including TENS, Hot pack and strengthening exercises will also be delivered along with Sacral Manipulation.
  Arms: Sacral Manipulation

SUMMARY:
* The study will be randomized clinical trial. This study will be conducted in University of Lahore Teaching Hospital, Lahore, Pakistan. A sample size of 84 will be randomly allocated into two experimental groups, (42 participants in each group), by lottery method. The participants, randomly allocated to the experimental group A, will receive Muscle Energy Technique (METs), Post isometric relaxation technique specifically, in addition with routine physical therapy as TENS, Hot pack, and strengthening exercises. METs will be performed on piriformis, iliopsoas, erector spine muscles, 1 set of 5 repetitions and 10 seconds hold.
* Participants in experimental group B, will get Sacroiliac joint manipulations with routine physical therapy by principal investigator.
* Both experimental groups will receive twelve treatment sessions and those will be given over a period of six weeks (2 sessions per week, each session of 30-40 minutes).
* Assessor will take outcome measures at baseline and at the end of 6th treatment week through Short Form McGill Pain Questionnaire, Roland-Morris Low Back Pain & Disability Questionnaire and Short Form Survey; SF-20.

DETAILED DESCRIPTION:
* Recruitment: Participants will be recruited and referred by orthopedic surgeon, University of Lahore Teaching Hospital to Physical Therapy Department.
* Screening: Diagnostic & pain provocative tests (Faber, Thigh thrust and Gillet tests) will be applied on recruited participants for screening. With all three positive tests, participants will be confirmed for positive SI joint dysfunction and will be considered eligible for entering the study.
* The FABER (Patrick's) Test stands for Flexion, Abduction and External Rotation. The participants will be positioned in supine. The leg will be placed in a figure-4 position (hip flexed and abducted with the lateral ankle resting on the contra-lateral thigh proximal to the knee. While stabilizing the opposite side of the pelvis at the anterior superior iliac spine, an external rotation, abduction and posterior force will be then lightly applied to the ipsilateral knee until the end range of motion would achieve. A further few small-amplitude oscillations would be applied to check for pain provocation at the end range of motion. A positive test will be the one that reproduces the participants' pain or limits their range of movement.
* Thigh thrust test is a posterior pelvic pain provocative test. It will be performed with the participant in supine lying, with the hip flexed to 90° (with bent knee) to stretch the posterior structures. By applying axial pressure along the length of the femur, the femur will be used as a lever to push the ilium posteriorly. One hand will be placed beneath the sacrum to fixate its position while the other hand will be used to apply a downward force to the femur. Broadhurst and Bond suggest adding hip adduction towards the mid line while Laslett & Williams advise to avoid excessive adduction due to discomfort for the participant. Test will be positive if it aggravates the pain in sacroiliac joint.
* The Stork test, also known as the Gillet Test, assesses the movement of the sacroiliac joint between the innominate and sacrum through the clinician's palpation, which may be a useful test for clinical evaluation of a subject's ability to stabilize intra-pelvic motion. The assessment of the Gillet's test involves palpation of the posterior superior iliac spine (PSIS). There are 2 phases to the Gillet's test: the stance phase and the hip flexion or swing phase. To perform this test, the patient will be asked to stand while the examiner will palpate the posterior superior iliac spine (PSIS) with one thumb and will palpate the base of the sacrum with the other thumb medial to the PSIS. The participants will be then instructed to stand on one leg while pulling the hip of the side being palpated into 90° or more of hip flexion. The test will then be repeated on the other side and compared bilaterally. The principal investigator will compare each side for quality and amplitude of movement. The test will be positive when the PSIS on the ipsilateral side (same side of the body) of the knee flexion move minimally in the inferior direction, doesn't move or is associated with pain. A positive test will be an indication of sacroiliac joint hypo-mobility.
* Randomization and Allocation: Afterwards, participants confirming the eligibility criteria will be randomly allocated, through lottery method, into two experimental groups (Group A, Group B).
* Blindness: Study will be single, assessor blinded and an independent investigator will perform randomization and will inform the patients and therapist about the allocation.
* Intervention: The participants, randomly allocated to the experimental group A, will receive METs (Post isometric relaxation technique specifically) in addition with routine physical therapy (TENS, Hot pack, and strengthening exercises). METs will be performed on piriformis, iliopsoas, erector spine muscles, 1 set of 5 repetitions and 10 seconds hold. Participants in experimental group B, will get Sacroiliac joint manipulations with routine physical therapy by principal investigator.
* Duration: Twelve treatment sessions will be given over a period of six weeks (2 sessions per week, each session of 30-40 minutes).
* Outcome Variables and Measures

  1. Pain (Short Form McGill Pain Questionnaire)
  2. Functional Disability (Roland-Morris Low Back Pain & Disability Questionnaire)
  3. Quality of Life (Short Form Survey; SF-20)
* Outcome measures will be taken at baseline and at the end of last treatment session i.e. 6th week. Collected data will be than analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diagnosed cases referred from orthopedic surgeon
* History of fall on buttock, lift and twist maneuver, overzealous kick
* Acute onset of sacral pain within period of 6 weeks
* FABER, Thigh thrust and Gillet sacral joint diagnostic tests must be positive to confirm the SI joint dysfunction before allocation

Exclusion Criteria:

* General low back pain, Sciatic pain, piriformis syndrome, Hip joint pathology
* SI joint spondylosis or ankylosing spondylitis
* Red flag signs positive (constant pain without movement, sudden weight loss with pain in time, lower limbs' undefined weakness, neurological signs)
* Structural leg length discrepancy and recent pregnancy
* Participants with other spinal pathologies (e.g. Osteomyelitis, Pott's disease, Cauda equine syndrome, spondylolisthesis or spondyloptosis, Lumbar disc herniation etc.)
* Participants with other systemic illnesses (e.g. cardiovascular disorders, gastrointestinal disorders, renal function disorders, Liver function disorders etc.)
* Participants with traumatic injuries (e.g. fractures, dislocations, sports injuries, road traffic accidents)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Short Form McGill Pain Questionnaire | 6 weeks
  Short form McGill Pain questionnaire (SF-MPQ 2) is 22-items, revised, short version and self-reported measure of pain. It assesses both the quality and intensity of subjective pain. It was initially developed by Dr. Melzack at McGill University in Montreal Canada. The four SF-MPQ-2 score ranges between 0 to 22 where o indicate no pain and 22 indicate worst possible pain.
Roland Morris disability and low back pain questionnaire | 6 weeks
  he Roland-Morris Questionnaire (RMQ) is a 24-items self-administered disability measure. Items would be scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24; higher scores will be represented as higher levels of pain-related disability.
Short Form Survey, SF-20 | 6 weeks
  The SF-20 is short version of SF-36 which is generic patient-reported outcome that qualifies health status and measures health related quality of life. The 20-Item Short Form Health Survey (SF-20) was developed in 1988 for the Medical Outcomes Study (MOS). In this scale, scores across each of its domains would be reported on a 0% to 100% scale, with 0% representing the worst possible score in that domain and 100% the best possible score. The exception to this scoring pattern would be the pain score, for which 0% will represent the best possible score and 100% the worst possible.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Sana Ashraf, MS-MSK*, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Telli H, Huner B, Kuru O. Determination of the Prevalence From Clinical Diagnosis of Sacroiliac Joint Dysfunction in Patients With Lumbar Disc Hernia and an Evaluation of the Effect of This Combination on Pain and Quality of Life. Spine (Phila Pa 1976). 2020 Apr 15;45(8):549-554. doi: 10.1097/BRS.0000000000003309. PMID 31842104
- [Background] Thawrani DP, Agabegi SS, Asghar F. Diagnosing Sacroiliac Joint Pain. J Am Acad Orthop Surg. 2019 Feb 1;27(3):85-93. doi: 10.5435/JAAOS-D-17-00132. PMID 30278010
- [Background] Orakifar N, Kamali F, Pirouzi S, Jamshidi F. Sacroiliac joint manipulation attenuates alpha-motoneuron activity in healthy women: a quasi-experimental study. Arch Phys Med Rehabil. 2012 Jan;93(1):56-61. doi: 10.1016/j.apmr.2011.05.027. PMID 22200384
- [Background] Garcia-Penalver UJ, Palop-Montoro MV, Manzano-Sanchez D. Effectiveness of the Muscle Energy Technique versus Osteopathic Manipulation in the Treatment of Sacroiliac Joint Dysfunction in Athletes. Int J Environ Res Public Health. 2020 Jun 22;17(12):4490. doi: 10.3390/ijerph17124490. PMID 32580480
- [Background] Zaidi F, Ahmed I. Effectiveness of muscle energy technique as compared to Maitland mobilisation for the treatment of chronic sacroiliac joint dysfunction. J Pak Med Assoc. 2020 Oct;70(10):1693-1697. doi: 10.5455/JPMA.43722. PMID 33159735
- [Background] de Toledo DFA, Kochem FB, Silva JG. High-velocity, low-amplitude manipulation (HVLA) does not alter three-dimensional position of sacroiliac joint in healthy men: A quasi-experimental study. J Bodyw Mov Ther. 2020 Jan;24(1):190-193. doi: 10.1016/j.jbmt.2019.05.020. Epub 2019 May 22. PMID 31987543
- [Background] Stratford PW, Riddle DL. A Roland Morris Disability Questionnaire Target Value to Distinguish between Functional and Dysfunctional States in People with Low Back Pain. Physiother Can. 2016;68(1):29-35. doi: 10.3138/ptc.2014-85. PMID 27504045
- [Background] Dworkin RH, Turk DC, Trudeau JJ, Benson C, Biondi DM, Katz NP, Kim M. Validation of the Short-form McGill Pain Questionnaire-2 (SF-MPQ-2) in acute low back pain. J Pain. 2015 Apr;16(4):357-66. doi: 10.1016/j.jpain.2015.01.012. Epub 2015 Jan 29. PMID 25640290
- [Background] Nejati P, Sartaj E, Imani F, Moeineddin R, Nejati L, Safavi M. Accuracy of the Diagnostic Tests of Sacroiliac Joint Dysfunction. J Chiropr Med. 2020 Mar;19(1):28-37. doi: 10.1016/j.jcm.2019.12.002. Epub 2020 Sep 12. PMID 33192189